CLINICAL TRIAL: NCT03628144
Title: The Use of Immunonutrition to Reduce Toxicities From Concurrent Chemotherapy and Radiotherapy for Treatment of Unresectable Stage IIIA-B Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Immunonutrition to Reduce Toxicities in Non-Small Cell Lung Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding unavailable
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Nestle Health Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MCC-19505
Record Dates: First submitted 2018-08-09; First posted 2018-08-14 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Non Small Cell Lung Cancer; NSCLC; Non-small Cell Lung Cancer; Non-small Cell Lung Cancer Stage IIIB; Non-small Cell Lung Cancer Stage ⅢA; NSCLC Stage IIIB; NSCLC, Stage IIIA
Keywords: Immunonutrition; Radiotherapy; Unresectable; Stage IIIA-B; Lung cancer; Radiation oncology; Thoracic oncology; Epidemiology; Nutrition
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Dietary Supplements; Radiotherapy; Drug Therapy; Standard of Care; Quality of Life; Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Randomized open-label, medical and radiation oncologist-blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- A: Intervention Group - Impact® (Experimental): A: Intervention Group - Standard of Care Concurrent Chemoradiotherapy (Chemotherapy + Radiation) with nutritional supplement. Impact® Advanced Recovery: Three times daily for the 5 days just prior to the start of each cycle of chemotherapy. Participants will undergo pre- and post-treatment assessments.
  Interventions: Dietary Supplement: Impact® Advanced Recovery; Radiation: Radiation Therapy; Drug: Chemotherapy; Other: Quality of life (EORTC-QLQ-30); Other: Evaluation of Cognitive Function (FACT-Cog, v. 3.0); Other: Mindfulness Questionnaire (FFMQ)
- B: Control Group - Boost® (Active Comparator): B: Control Group - Standard of Care Concurrent Chemoradiotherapy (Chemotherapy + Radiation) with nutritional supplement. Boost® High Protein: Identical schedule of a supplement with similar calorie and protein content, Boost® High Protein. Participants will undergo pre- and post-treatment assessments.
  Interventions: Dietary Supplement: Boost® High Protein; Radiation: Radiation Therapy; Drug: Chemotherapy; Other: Quality of life (EORTC-QLQ-30); Other: Evaluation of Cognitive Function (FACT-Cog, v. 3.0); Other: Mindfulness Questionnaire (FFMQ)

INTERVENTIONS:
Dietary Supplement: Impact® Advanced Recovery — The intervention drink Impact® will be ingested every two weeks since usually chemotherapy is delivered concurrently with radiation therapy in 2 week cycles. For patients who are placed on weekly or every 4 weeks chemotherapy dosing schedules, the treatment and control supplements will still be given every two weeks.
  Other Names: Nutritional supplement
  Arms: A: Intervention Group - Impact®
Dietary Supplement: Boost® High Protein — The control supplement drink Boost® will be ingested every two weeks since usually chemotherapy is delivered concurrently with radiation therapy in 2 week cycles. For patients who are placed on weekly or every 4 weeks chemotherapy dosing schedules, the treatment and control supplements will still be given every two weeks.
  Other Names: Nutritional supplement
  Arms: B: Control Group - Boost®
Radiation: Radiation Therapy — Standard of Care: Weekly radiation therapy as already planned for each participant, at Moffitt clinic visits.
  Other Names: Radiotherapy
Drug: Chemotherapy — Standard of Care: Chemotherapy as already planned for each participant.
  Other Names: Standard of Care
Other: Quality of life (EORTC-QLQ-30) — Participants will undergo pre- and post-treatment assessments.
  Other Names: Questionnaire
Other: Evaluation of Cognitive Function (FACT-Cog, v. 3.0) — Participants will undergo pre- and post-treatment assessments.
  Other Names: Questionnaire
Other: Mindfulness Questionnaire (FFMQ) — Participants will undergo pre- and post-treatment assessments.
  Other Names: Questionnaire

SUMMARY:
The purpose of this study is to assess whether either or both nutrition supplements (Impact® Advanced Recovery or Boost® High Protein) ingested prior to and during concurrent chemoradiotherapy decreases toxic side effects of treatment in Stage IIIA-B non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be recruited from the Moffitt Cancer Center Thoracic Oncology Outpatient Clinic when identified by a thoracic oncologist that the patient will undergo all of their chemoradiotherapy at Moffitt.

  * Men and women ≥18 years of age.
  * Diagnosed with unresectable stage IIIA or IIIB non-small cell lung cancer.
  * Patients plan to undergo all cancer treatment at Moffitt Cancer Center with definitive concurrent chemotherapy and radiotherapy.
  * No prior treatment of NSCLC.
  * Able to provide informed consent.
  * Performance status 0, 1 or 2.
  * Life expectancy >3 months.
  * No esophagitis within 90 days.

Exclusion Criteria:

* Mental incompetence or chronic psychiatric disease.
* Incarcerated individuals.
* Use of antibiotics or probiotic supplements within one month of chemoradiotherapy.
* Allergy to any of the components of Impact® Advanced Recovery or Boost® High Protein.
* Pregnant female or breast-feeding. Any female patient <45 years old not using appropriate contraceptive measures during the treatment.
* Sepsis or active infection.
* Chronic renal failure stage IV (requiring protein restriction) or stage V requiring dialysis.
* Malnutrition defined as BMI <16.
* Inflammatory bowel disease (ulcerative colitis or Crohn's disease).
* Severe hepatic dysfunction (baseline prothrombin time off any anticoagulation of international normalized ratio (INR) >1.8).
* Significant digestive disease with nausea, vomiting or diarrhea, NCI Grade >1.
* Use of IL-6 inhibitors (tocilizumab or siltuximab) within last 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-07 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment Related Adverse Events Per Study Arm | Up to 48 months
  Overall toxicity from therapy as assessed by NCI Common Toxicity Criteria for Adverse Events (CTCAE) v. 5.0 that directly correlates with toxicity from concurrent chemoradiotherapy. Based on another randomized trial using pretreatment immunonutrition, investigators want to see if this nutritional intervention will likely decrease overall chemoradiotherapy related toxicity. All toxicity and adverse events (CTCAE v.5.0) will be assessed weekly and attributed by the treating radiation oncologist and entered into the clinical trials management database OnCore for later statistical analysis. Differences in toxicity events at the end of the study in participants receiving Impact® and those receiving Boost® will be compared using two-sample t-test.
Change in Plasma Levels of IL-6 Per Study Arm | Up to 48 months
  Measurement of the marked change of IL-6 that directly correlates with toxicity from concurrent chemoradiotherapy. Multiplex immunoassay will be used to determine the plasma levels of IL-6 in pg/ml as a continuous variable. Two-sample t-test for change in IL-6 at the last visit from the baseline will be compared between the two arms. Kolmogorove-Smirnov and Jarque-Bera tests will be performed to test for normality assumption on the primary endpoints prior to t-test analysis. If either test indicates a violation of the normality assumption, investigators will use an appropriate rank-based Wilcoxon rank-sum test instead of t-test.

SECONDARY OUTCOMES:
Overall Survival (OS) 9OS) | Up to 2 years
  Overall survival (OS) defined as the length of time interval between the date of cancer treatment completion and the date of death due to any cause. Kaplan-Meier curves will be estimated for each arm. Log-rank test will be performed to examine the effect of Impact® vs. Boost® on measures of OS.
Progression-free Survival (PFS) | Up to 2 years
  Progression-free survival (PFS) will be assessed using the length of time interval from the cancer treatment completion to the earlier of the first documentation of disease progression or death from any cause. Kaplan-Meier curves will be estimated for each arm. Log-rank test will be performed to examine the effect of Impact® vs. Boost® on measures of PFS.
Rate of Treatment Changes or Interruptions Per Study Arm | Up to 2 years
  Treatment interruptions, chemotherapy dose reduction or hospitalizations secondary to toxicity.
Rate of Participant Regimen Compliance Per Study Arm | Up to 2 years
  Rate of participant compliance, with immunonutrition regimen, according to participant diaries. Each participant will complete a compliance diary noting when each carton/bottle of the study agent is drunk and the card will be collected by the Study Coordinator at on treatment clinic visits (OTV) prior to receiving the new batch of study or control supplements.

CONTACTS AND LOCATIONS:
Overall Officials: Lary A. Robinson, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States